CLINICAL TRIAL: NCT04737876
Title: A Phase 1, Randomized, Single-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Fecal Pharmacokinetics of Orally Administered BX002-A in Healthy Adult Individuals
Brief Title: A Study to Evaluate the Safety, Tolerability, and Fecal Pharmacokinetics of BX002-A in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BiomX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BMX-02-001
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BX002-A (Experimental): BX002-A: 1 mL liquid for multiple dose oral administration
  Interventions: Biological: BX002-A
- Placebo (Placebo Comparator): Placebo: 1 mL liquid for multiple dose oral administration
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BX002-A — bacteriophage cocktail
  Arms: BX002-A
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of study BMX-02-001 is to evaluate the safety, tolerability and feasibility of orally administered BX002-A to deliver viable bacteriophages to the gut.

DETAILED DESCRIPTION:
Study BMX-02-001 is a randomized, single-blind, placebo-controlled study to evaluate the safety, tolerability, and feasibility of orally administered BX002-A to deliver viable phages that can be measured in the stool.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18-65 years old
2. Able to understand study procedures and sign informed consent

Exclusion Criteria:

1. Evidence or history of clinically significant underlying conditions
2. Women who are pregnant or nursing, or plan to become pregnant during study, or women of childbearing potential not using adequate contraceptive measures
3. History of constipation, severe diarrhea and/or loose stools within 14 days
4. History of procedures aimed at modifying the gastrointestinal microbiota within past year (e.g., fecal microbiota transplantation)
5. Topical gastrointestinal treatment (e.g., enemas) in the 2 weeks prior or planned during study
6. Use of bowel cleansing or preparation in the 4 weeks prior or planned during study
7. Participation in another investigational trial within 30 days
8. Known allergy or hypersensitivity to an excipient in the study drug or placebo
9. Any other reason which according to investigator may impact proper study conduct
10. History of alcohol abuse; drug or medication abuse or tobacco use
11. Subject who cannot be contacted in case of emergency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: adverse events | Through study completion Day 31 (+ 2 days)
  Evaluated by reviewing adverse events

OTHER OUTCOMES:
Plaque-Forming Unit analysis | Day -1 through Day 6
  Quantitative measurement of viable phage in stool after oral administration of BX002-A via plaque-forming unit analysis

CONTACTS AND LOCATIONS:
Overall Officials: Physician, Study Director — BiomX, Inc.
Locations (1):
- Medical Facility, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No